CLINICAL TRIAL: NCT01579552
Title: EMPOWER Study: Promoting Breast Cancer Screening in Women Who Survived Childhood Cancer
Brief Title: Promoting Breast Cancer Screening in Women Who Survived Childhood Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: St. Jude Children's Research Hospital (Other); University of Colorado, Denver (Other); Dana-Farber Cancer Institute (Other); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-104
Record Dates: First submitted 2012-04-03; First posted 2012-04-18 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Questionnaires; telephone counseling session; 10-104; Childhood Cancer Survivor Women Post Chest Radiation
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

ARMS (2):
- Intervention Group (Experimental): The EMPOWER intervention trial is a 12-month study of 360 women from the Childhood Cancer Survivor Study who have previously been treated with chest radiation, are 25 to 49 years of age at the time of enrollment, are 8 years or more since their chest radiation, and have not had a mammogram or other breast imaging study in the preceding two years. Following a baseline questionnaire, participants will be randomized to the attention control group (N=120) or the intervention group (N=240).
  Interventions: Behavioral: survey, questionaire
- attention control group (Active Comparator): The EMPOWER intervention trial is a 12-month study of 360 women from the Childhood Cancer Survivor Study who have previously been treated with chest radiation, are 25 to 49 years of age at the time of enrollment, are 8 years or more since their chest radiation, and have not had a mammogram or other breast imaging study in the preceding two years. Following a baseline questionnaire, participants will be randomized to the attention control group (N=120) or the intervention group (N=240).
  Interventions: Behavioral: survey, questionaire

INTERVENTIONS:
Behavioral: survey, questionaire — The intervention components (mailed tailored print materials followed by telephone-delivered Brief MI). Following enrollment into the study and completion of the informed consent form and baseline survey, participants will be randomized to the active intervention group or the attention control group. The data that will be used in the analysis will come from the baseline survey, medical records of breast imaging studies, and a 12-month follow-up questionnaire.
  Arms: Intervention Group
Behavioral: survey, questionaire — The intervention components (mailed tailored print materials followed by telephone-delivered Brief MI). Following enrollment into the study and completion of the informed consent form and baseline survey, participants will be randomized to the active intervention group or the attention control group. The data that will be used in the analysis will come from the baseline survey, medical records of breast imaging studies, and a 12-month follow-up questionnaire.
  Arms: attention control group

SUMMARY:
The purpose of this study is to empower women to improve their health in two very important areas: breast and heart health. This twelve-month study will compare two methods of informing participants about potential health risks and ways to stay healthy.

The EMPOWER Study has been designed for adult women who were treated for a childhood cancer with chest radiation.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the CCSS cohort
* Diagnosed with a childhood cancer prior to 21 years of age
* Treated with > 20 Gy of chest radiation (mantle, mediastinal, lung, or chest)
* Age 25-49 years at time of enrollment into the study
* Interval from chest radiation to the time of enrollment of > 8 years
* No mammogram or other breast imaging study in the 24 months prior to enrollment
* English-speaking - The University of Colorado AMC Denver and MSKCC group are not capable of or equipped for conducting a brief motivational interviews by telephone in another language.

Exclusion Criteria:

* Diagnosed with breast cancer
* Participated in the Project VISION feasibility study (exposed to part of the intervention)

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
efficacy | 12 months
  Determine the efficacy of an intervention, consisting of mailed tailored print materials followed by a telephone-delivered Brief Motivational Interview, on mammogram screening rates compared with an attention control. Mammogram completed by 12-month questionnaire (confirmed by medical record)

SECONDARY OUTCOMES:
Moderating factors | 12 months
  By including interaction terms in the model, we will assess potential moderating factors such as age, race/ethnicity, health insurance, & other sociodemographic variables. Moderating effects can be adequately addressed through interactions between the intervention & the above mentioned covariates.124 An interaction with the treatment group indicator suggests differential effectiveness, and moderator variables with statistically significant interactions will remain in the model. Interactions will be estimated using crossproduct terms between the intervention indicator & the mediating variable.
Mediating factors | 12 months
  Based on results from the MPS & breast ca screening intervention trials among women in the general pop or familial risk, we are a priori interested in mediating effect of 5 variable domains: knowledge of screening guidelines, breast ca health beliefs, decisional balance of the pros & cons of mammography, self-efficacy, & psychological factors. For each of these domains, a global or subscale score will be used as appropriate. For ex, from the BSI-18, a global score of psychological symptoms & a subscale score for each group of symptoms can be estimated.
Economic analysis | 12 months
  Replication costs of intervention: dollar cost; time cost (per person)
  • Costs resulting from intervention: total cost of screening/diagnostic imaging, diagnostic procedures, breast surgery, non-procedure breast-related physician visits
Breast MRI completed by 12-month questionnaire | 12 months
  (confirmed by medical record)
  • Barriers to completing breast MRI: moderating/mediating variables listed above

CONTACTS AND LOCATIONS:
Overall Officials: Chaya Moskowitz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Oeffinger KC, Ford JS, Moskowitz CS, Chou JF, Henderson TO, Hudson MM, Diller L, McDonald A, Ford J, Mubdi NZ, Rinehart D, Vukadinovich C, Gibson TM, Anderson N, Elkin EB, Garrett K, Rebull M, Leisenring W, Robison LL, Armstrong GT. Promoting Breast Cancer Surveillance: The EMPOWER Study, a Randomized Clinical Trial in the Childhood Cancer Survivor Study. J Clin Oncol. 2019 Aug 20;37(24):2131-2140. doi: 10.1200/JCO.19.00547. Epub 2019 Jul 1. PMID 31260642
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/